CLINICAL TRIAL: NCT00195546
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled Study of DVS-233 SR for Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating DVS-233 SR for Treatment of Vasomotor Symptoms Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A2-321
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Menopause
Keywords: Menopause

INTERVENTIONS:
Drug: DVS-233

SUMMARY:
Primary: To assess the efficacy and safety of DVS-233 SR compared with placebo for treatment of vasomotor symptoms (VMS) associated with menopause and to compare the bleeding incidence of DVS-233 SR and tibolone. Secondary: To assess the effects of DVS-233 SR and tibolone on changes from baseline in weight, breast pain, and health outcomes indicators.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women of age 40 to 65 seeking treatment for hot flashes with last natural menstrual period (LNMP) completed at least 12 months prior to screening.
* Minimum of 7 moderate to severe hot flashes per day or 50 per week recorded for 7 consecutive days
* Body Mass Index less than or equal to 34 kg/m2 using the nomograph for BMI.

Exclusion Criteria:

* History, presence, or suspicion of estrogen-dependent neoplasia; Malignancy, or treatment for malignancy, within the previous 2 years.
* Active or recent arterial thromboembolic disease; History of venous thromboembolism
* History of cerebrovascular accident, stroke, or transient ischemic attack -
* Presence of major depressive disorder, bipolar disorder, psychotic disorder, or generalized anxiety disorder requiring therapy
* Persistent elevated blood pressure

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2005-04; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of DVS-233 SR compared with placebo for treatment of vasomotor symptoms (VMS) associated with menopause and to compare the bleeding incidence of DVS-233 SR and tibolone.

SECONDARY OUTCOMES:
To assess the effects of DVS-233 SR and tibolone on changes from baseline in weight, breast pain, and health outcomes indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Finland, Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Ukraine, Romania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Czech Republic, WPPGCLI@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Hungary, Croatia, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Poland, WVWZMED@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezlj@wyeth.com
Locations (35):
- Leuven, Belgium
- Croatia (2):
  - Zadar
  - Zagreb
- Czechia (3):
  - Olomuc
  - Ostrava
  - Přerov
- Finland (2):
  - Kuopio
  - Oulu
- France (2):
  - Évry
  - Paris
- Hungary (2):
  - Debrecen
  - Tatabánya
- Mexico (2):
  - Del. Cuauhtemoc
  - Lomas Virrteyes
- Netherlands (3):
  - 's-Hertogenbosch
  - Hengelo
  - Nijmegen
- Poland (4):
  - Katowice
  - Poznan
  - Warsaw
  - Wroclaw
- Bucharest, Romania
- South Africa (3):
  - Bloemfontein
  - Centurion
  - Parow
- Madrid, Spain
- Sweden (3):
  - Linköping
  - Stockholm
  - Uppsala
- Ukraine (2):
  - Donetsk
  - Kyiv
- United Kingdom (4):
  - Fowey
  - Leicester
  - London
  - Plymouth